CLINICAL TRIAL: NCT05406791
Title: Technology Enabled Services to Enhance Depression Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Rush University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Mohr, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU#:00211887; 1P50MH119029-01A1 (NIH)
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensor-enabled digital mental health intervention (DMHI) (Experimental): Patients randomized to sensor-enabled DMHI condition will use Ksana Health's "Vira" mobile therapy platform with support from a study coach
  Interventions: Other: VIRA App
- Experimental: Control Treatment (CT) (Experimental): Participants randomized to the CT condition will use a Mood Education App designed by researchers at the University of Virginia to deliver psychoeducational content to help people self-manage symptoms of depression, anxiety, and stress.
  Interventions: Other: Mood Education App

INTERVENTIONS:
Other: VIRA App — Support from coach and using the VIRA app
  Arms: Sensor-enabled digital mental health intervention (DMHI)
Other: Mood Education App — Support from mood education app
  Arms: Experimental: Control Treatment (CT)

SUMMARY:
This study will compare two digital mental health interventions (DMHIs). One DMHI will use an app called Vira (which is a product developed and managed by Ksana Health), along with low intensity coaching provided via phone and both SMS text and in-app messaging. The other DMHI will provide a broad range of information on how to manage symptoms of depression, anxiety, and stress. The DMHI will be evaluated with patients receiving care from Rush University Medical Center's primary care and family medicine clinics, which serve racially, ethnically, and economically diverse communities; evaluations may also be extended beyond Rush patients.

DETAILED DESCRIPTION:
Depression and anxiety are common and impose a tremendous societal burden in terms of cost, morbidity, quality of life, and mortality. Yet, few people are able to obtain adequate or appropriate treatment.

This trial will compare the ability of two digital mental health interventions (DMHIs) to reduce depression and anxiety. One DMHI, called Mood Education App, provides information on depression and a broad range of strategies that are effective in improving symptoms. The other app, called VIRA, uses smartphone sensors to identify a few behavioral markers, including mobility patterns, physical activity, and sleep. The results of these sensed behavioral markers are used to give the participant behavior change recommendations through the Vira app that are expected to result in symptom improvement. The DMHI will include low intensity coaching, which includes one or more brief phone calls and communication via SMS text and in-app messaging. Both treatments are 8-weeks long.

The trial will be conducted within Rush University Medical Center's primary care and family medicine clinics, although recruitment be expanded beyond these clinics.

ELIGIBILITY:
Inclusion Criteria:

* US Citizen/ Resident
* 13 years or older
* English Speaking
* Owns an Android or iPhone smartphone with an up-to-date operating system
* Has used a smartphone in the last 7 days
* PHQ-8 greater than or equal to 10 and/or GAD-7 greater than or equal to 10

Exclusion Criteria:

* Children under the age of 13
* Severe suicidality (as defined by presence of a plan + intent to act on that plan)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Mohr, PhD, Principal Investigator — Northwestern University
Locations (1):
- Rush University Medical Center Department of Psychiatry & Behavioral Sciences, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the NIMH Data Archive
Time Frame: Data will be available 1 year after completion of the study.
Access Criteria: Approval by NIMH Data Archive
URL: https://nda.nih.gov/

REFERENCES:
- [Derived] Stiles-Shields C, Reyes KM, Lakhtakia T, Smith SR, Barnas OE, Gray EL, Krause CJ, Kruzan KP, Kwasny MJ, Mir Z, Panjwani S, Rothschild SK, Sanchez-Johnsen L, Winquist NW, Lattie EG, Allen NB, Reddy M, Mohr DC. A personal sensing technology enabled service versus a digital psychoeducation control for primary care patients with depression and anxiety: a pilot randomized controlled trial. BMC Psychiatry. 2024 Nov 19;24(1):828. doi: 10.1186/s12888-024-06284-z. PMID 39563248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between June 2022 and June 2023. Patients were recruited in-person from clinic-based sites and through community events (e.g., back-to-school fairs, wellness events); the electronic health record (EHR; MyChart/Epic); social media and other platforms; and through subject recruitment registries.
Pre-assignment Details: Of 258 individuals assessed for eligibility, 130 met inclusion criteria and were randomized to treatment groups.
Period: Overall Study
Arm/Group | Sensor-enabled Digital Mental Health Intervention (DMHI) | Experimental: Control Treatment (CT)
Started | 65 | 65
Completed | 52 | 55
Not Completed | 13 | 10
Not completed — Lost to Follow-up | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensor-enabled Digital Mental Health Intervention (DMHI) | Experimental: Control Treatment (CT) | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 62 | 62 | 124
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [25 to 38] | 33 [26 to 40] | 32 [25 to 39]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 52 | 49 | 101
  Male | 12 | 12 | 24
  Non-binary | 0 | 4 | 4
  Transgender | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 53 | 53 | 106
    Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 16 | 28
  Not Hispanic or Latino | 53 | 48 | 101
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 15 | 33
  White | 35 | 33 | 68
  More than one race | 6 | 9 | 15
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 65 | 65 | 130
Education [Count of Participants; unit: Participants]
  Some high school or less | 4 | 3 | 7
  High School Graduate/ GED | 6 | 5 | 11
  Vocational/Technical Degree, Associate's Degree, or Some College | 18 | 15 | 33
  Bachelor's Degree | 18 | 17 | 35
  Post-Bachelors Education | 19 | 24 | 43
  Prefer not to answer | 0 | 1 | 1
Marital Status [Count of Participants; unit: Participants]
  Divorced | 2 | 0 | 2
  Living with Partner | 8 | 10 | 18
  Married | 17 | 15 | 32
  Separated | 0 | 2 | 2
  Single | 37 | 37 | 74
  Widowed | 1 | 1 | 2
Household Income [Count of Participants; unit: Participants]
  Less than $10,000 | 6 | 3 | 9
  $10,000 - $19,999 | 4 | 9 | 13
  $20,000 - $39,999 | 7 | 5 | 12
  $40,000 - $59,999 | 7 | 2 | 9
  $60,000 - $99,999 | 14 | 14 | 28
  $100,000 + | 20 | 23 | 43
  Don't know | 4 | 6 | 10
  Prefer not to answer | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionaire-9 (PHQ-9)
Description: The PHQ-9 measures depression symptom severity on a scale of 0-27, with higher scores indicating greater symptom severity.
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sensor-enabled Digital Mental Health Intervention (DMHI) | Experimental: Control Treatment (CT)
Number analyzed (Participants) | 65 | 65
score on a scale
  Baseline | 13.2 [11.6 to 14.8] | 12.4 [10.8 to 14.0]
  Week 4 | 10.0 [8.3 to 11.6] | 9.4 [7.8 to 11.1]
  Week 8 | 9.5 [7.8 to 11.2] | 9.2 [7.6 to 10.8]
  Week 12 | 8.7 [6.8 to 10.5] | 7.9 [6.2 to 9.5]

2. Primary Outcome: Generalized Anxiety Disorder-7 (GAD-7)
Description: The GAD-7 measures anxiety symptom severity on a scale of 0-21, with higher scores indicating greater symptoms severity
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sensor-enabled Digital Mental Health Intervention (DMHI) | Experimental: Control Treatment (CT)
Number analyzed (Participants) | 65 | 65
score on a scale
  Baseline | 11.7 [10.2 to 13.2] | 12.2 [10.7 to 13.7]
  Week 4 | 8.8 [7.3 to 10.3] | 9.8 [8.3 to 11.3]
  Week 8 | 8.2 [6.5 to 9.9] | 9.3 [7.8 to 11.0]
  Week 12 | 7.5 [5.7 to 9.4] | 7.4 [5.9 to 9.0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 12 weeks
Description: Adverse events were monitored via assessments completed by participants (completed by all arms), application user feedback interviews (intervention arm-only), and interactions with the coaches (intervention arm-only). Questions regarding suicidal ideation were explicitly asked only on assessment questions (PHQ-9). The open-ended nature of interviews and coach interaction allowed for expression of suicidal thoughts or behaviors and as a result was monitored for indications of adverse events.
Arm/Group | Sensor-enabled Digital Mental Health Intervention (DMHI) | Experimental: Control Treatment (CT)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT05406791/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT05406791/SAP_001.pdf
  • Informed Consent Form (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT05406791/ICF_002.pdf